CLINICAL TRIAL: NCT05171738
Title: Appraisal of Two Different Approaches of Micro-osteoperforations During Maxillary Molar Distalization Via Skeletally-anchored Distaljet Appliance
Brief Title: Distalization Via Skeletally-anchored Distaljet Appliance With Two Approaches of Micro-osteoperforations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, khaled abd el khaliq hendy, BDS (2017), Faculty of Dental Medicine (Cairo-Boys) Al-Azhar University, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 788/309
Record Dates: First submitted 2021-11-29; First posted 2021-12-29 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Class II Division 1 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group(1) (Active Comparator): Group I: will include ten patients undergo maxillary molar distalization using skeletally anchored distal jet appliance with MOPs that will be performed buccally on repeated basis on two sides before and during maxillary molar distalization
  Interventions: Device: skeletally anchored distal jet
- group(2) (Active Comparator): Group II:will include ten patients undergo maxillary molar distalization using skeletally anchored distal jet appliance with MOPs that will be performed both buccally and palatally on repeated basis on two sides before and during maxillary molar distalization.
  Interventions: Device: skeletally anchored distal jet

INTERVENTIONS:
Device: skeletally anchored distal jet — used from day one and activated every month

SUMMARY:
study will be directed to evaluate two approaches of micro-osteoperforations during maxillary molar distalization.

DETAILED DESCRIPTION:
Maxillary molar distalization via skeletally anchored distal jet appliance randomly divided into two equal groups

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

All patients should satisfy the following criteria:-

1. Age range from 13-17 years.
2. Bilateral Class II molar relationship.
3. Skeletal Class I or mild Class II relationship.
4. Normodivergent skeletal pattern
5. No posterior crowding or diastemas.
6. Fully erupted maxillary first and second molars.
7. Congenitally missing or extracted third molars.
8. Good oral and general health.
9. No systemic disease/medication that could interfere with OTM.
10. No previous orthodontic treatment.

Exclusion Criteria:

* Exclusion criteria:

  1. Patient diagnosed to have an indication for non-extraction approach.
  2. Poor oral hygiene or periodontally compromised patient.
  3. Patient with craniofacial anomalies or previous history of trauma, bruxism or parafunctions.
  4. Previous orthodontic treatment

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
change in molar postion | from start of treatment until study completion, an average of 1 year
  using cephalometric x_ray for measurment

CONTACTS AND LOCATIONS:
Locations (1):
- Al azhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided